CLINICAL TRIAL: NCT06945133
Title: Correlation Study Between the Classification of Arthrogenic Motor Inhibition (AMI) and Clinical Assessment After ACL Rupture
Acronym: AMIVAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A00125-44; 2025-A00125-44 (Other: ANSM)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMI testing group (Experimental): Interventions administered are the following :
  * Surface EMG to measure inhibition of the VM and the RF on the injured and non-injured sides during attempts at voluntary contractions of the knee extensor muscles.
  * Myotonometry to measure the stiffness of the semi-membranosus and biceps femoris (long head) on the injured and non-injured sides under resting conditions
  Interventions: Other: Clinical testing

INTERVENTIONS:
Other: Clinical testing — Intervention includes :
  * Surface EMG to measure inhibition of the VM and the rectus femoris (RF) on the injured and non-injured sides during attempts at voluntary contractions of the knee extensor muscles.
  * Myotonometry to measure the stiffness of the semimembranosus and biceps femoris (long head) on the injured and non-injured sides under resting conditions

SUMMARY:
The goal of this interventional study is to measure medial vastus inhibition and associate it with AMI classification in patients with ACL rupture. The main question it aims to answer is:

Is there a correlation between AMI classification and clinical assessment after ACL rupture ? Participants will undergo surface EMG and Myotonometry.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years and < 45 years
* Patient with an ACL rupture confirmed by MRI
* Patient with an ACL rupture ≤ 30 days old
* French speaking patient who does not object to the use of his/her data

Exclusion Criteria:

* Patient with previous ipsi or contralateral knee injury/surgery
* Patient with multi-ligament injury
* Pregnant or breastfeeding woman

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Surface EMG and AMI correlation | From enrollment to Day 30
  Electrical signal amplitude, expressed in mV, is evaluated at the level of the VM. This electrical signal amplitude is correlated with the level of muscle activation. It is measured with a surface EMG, which measures the activation of the VM during a voluntary attempt to contract the knee extensors. The ratio: Amplitude of the electrical signal from the injured side of the VM / Amplitude of the electrical signal from the non-injured side of the VM is used to determine the inhibition of the VM.
  AMI is assessed using the Sonnery-Cottet classification (Sonnery-Cottet et al, 2022)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No